CLINICAL TRIAL: NCT03239925
Title: Acute Effects of Cell Phone Exposure on Immediate Attention Levels and Concentration of Emergency Physicians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karadeniz Technical University (Other)
Collaborators: Trabzon Kanuni Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Suleyman Turedi, Prof. MD., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-49
Record Dates: First submitted 2017-07-24; First posted 2017-08-04 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Acute Effects of EMWs Emitted by Cell Phones
Keywords: Cell phones, Electromagnetic Radiation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental group: we planned that all participants in this group would hold a cell phone to their left ears in their left hands, in 'on' mode, for 15 min, and that they would thus be exposed to a 900-1800 MHz magnetic field (EMW) for 15 min.
  Control group: these would hold a cell phone to their left ears in their left hands for 15 min in 'off' mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): all participants in this group would hold a cell phone to their left ears in their left hands, in 'on' mode, for 15 min, and that they would thus be exposed to a 900-1800 MHz magnetic field (EMW) for 15 min.
  Interventions: Radiation: Electromagnetic field of cell phone in ''on'' mode.
- Control group (Placebo Comparator): these would hold a cell phone to their left ears in their left hands for 15 min in 'off' mode
  Interventions: Radiation: Electromagnetic field of cell phone in 'off' mode.

INTERVENTIONS:
Radiation: Electromagnetic field of cell phone in ''on'' mode. — In experimental group, participants would hold a cell phone to their left ears in their left hands, in 'on' mode, for 15 min, and that they would thus be exposed to a 900-1800 MHz magnetic field (EMW) for 15 min.
  Other Names: Experimental group
  Arms: Experimental group
Radiation: Electromagnetic field of cell phone in 'off' mode. — In control group, participants would hold a cell phone to their left ears in their left hands for 15 min in 'off' mode.
  Other Names: Control group
  Arms: Control group

SUMMARY:
To investigate the acute effects of cell phone exposure on immediate attention levels and concentration of emergency department physicians

DETAILED DESCRIPTION:
The development of new media technologies has made these an indispensible part of human life. Increasing cell phone use is to a large extent a component of this development.

The effects on humans of electromagnetic waves (EMW) has been a subject of particular interest and concern in recent years.

Cell phone technology; With the Wireless Local Area Network (WLAN), Bluetooth and Digital Enhanced Cordless Telecommunications (DECT), cell phones have become one of the most commonly used sources of EMW to which humans are today exposed.

Concerns over the effects of EMW (at a range of 900-1800 MHz) cell phone receivers may be associated with carcinogenic and neuronal activity. Excessive use of cell phones is known to cause headache, a feeling of discomfort and a warm sensation around the ear. In addition, it is thought to have side-effects including memory loss, depression and adverse impacts on attention and concentration.

Attention is defined as the individual directing his mental receptors toward a stimulus or stimuli occurring in the phenomenal environment, of which he is aware and which he can perceive with his sense organs. Attention is also a nervous system function permitting the individual to concern himself solely with stimuli in the context of needs and aims at that moment from among the many stimuli in the environment.

One of the significant features of attention is that it is selective. There are many stimuli around us potentially capable of attracting our attention. Since it is impossible to focus on all of these, one must be able to select the important ones. Selective attention refers to the ignoring of other stimuli by identifying the important one and directing one's attention to a specific stimulus. In other words, it means reacting only to relevant stimuli, not to irrelevant ones.

Emergency care means the prompt provision of the medical care required by an individual with a life-threatening condition. Emergency departments are units that provide this service for patients requiring emergency care. Emergency departments are places in which health personnel are in a constant state of activity and have to provide constant services at an intense work rate. Personnel such as emergency medicine specialists and emergency medicine assistant physicians or other specialist physicians and practitioners, nurses, health administrators, emergency medicine technicians and ancillary staff work in emergency departments. Emergency department personnel are exposed to very significant stress factors, such as taking immediate and vitally important decisions, an intense work rate, long shifts, insufficient rest time, and the need to cope with rude and aggressive patients and relatives. These stress factors are estimated to affect health workers' attention levels, decision-making abilities and concentration. Factors such as inattention and memory errors that compromise that compromise the individual's concentration are reported to pay an important role in medical errors in emergency departments. The importance of attention and concentration is obvious in emergency departments, where vital decisions are made concurrently, and where medical procedures must be performed to perfection and in a race against time. Combatting factors that have a negative impact on this is highly important. The hypothesis that cell phones and electromagnetic fields may have an effect on this attention and concentration constituted the basis of the current study.

Cell phone use among emergency department physicians is widespread, as in all other fields. Cell phone use is particularly important for requesting consultations in patient management in the emergency department.

The purpose of this study is to investigate the acute effects on emergency physicians' attention and concentration of EMWs emitted by cell phones.

Study protocol

At the beginning of the study, emergency department physicians were asked to complete an assessment form in order to determine the inclusion and exclusion criteria (App-1).

The investigators were planned to enroll 30 emergency physicians on the basis of the inclusion and exclusion criteria described above.

An internet-based power analysis program was used to calculate the sample size (UCSF Biostatistics:Power and sample size programs. http://www.biostat.ucsf.edu/sampsize.html#G*Power.) According to a preliminary study the investigators were performed before EMW exposure, emergency physicians' mean attention level was determined at 75. The sample size was calculated predicting a 50% decrease with EMW exposure. The investigators were therefore targeted 30 participants, 15 in each group, for 80% power.

The investigators were planned to apply the d2 test of attention, which is widely recognized in the literature, to assess attention and concentration before the study, to all the physicians enrolled. Based on TN-E scores in the d2 test of attention, the participants were listed in order of highest score to lowest. Following that procedure, two-way randomization was applied and two groups (experimental and control) with similar initial attention level were established using the head-tail method.

Experimental group: The investigators were planned that all participants in this group would hold a cell phone to their left ears in their left hands, in 'on' mode, for 15 min, and that they would thus be exposed to a 900-1800 MHz magnetic field (EMW) for 15 min.

Control group: these would hold a cell phone to their left ears in their left hands for 15 min in 'off' mode.

Throughout the study, The investigators were planned that the cell phone screen would be covered with black tape, and that all participants and the author performing subsequent attention evaluations would be unaware whether the cell phone was 'on' or 'off'.

Following this 15-min procedure, The investigators were planned that the d2 test of attention would be administered to both groups by a specialist psychologist in a blinded manner, and planned to compare attention and concentration levels between the experimental group exposed to EMW via cell phone and the non-exposed control group.

d2 test of attention: A time-dependent test measuring selective attention and concentration. Other parameters measured are speed of performance, rule compliance and performance quality. The test can be administered individually or in groups between the ages of 9 and 60. The test form contains 14 rows with 47 figures in each. The letters 'd' and 'p' are used in the test. Up to four marks are placed above, below or both above and below some letters. There are 16 total possible forms, depending on the marks on the letters.

The task of the person administered the test is to find all the letters 'd' with two marks. The subject is allowed 20 seconds to complete the task set out in each row and is asked to find all the letters 'd' with two marks. The test takes approximately 8 min to administer. Evaluation of the test is based on TN: Total number of symbols marked (psycho-motor speed), E1: Number of symbols skipped without being marked (selective attention), E2: Number of symbols marked incorrectly (special learning difficulty), E: Focusing level, CP: Total number of correct marks , TN-E: Total number of items minus error score (test performance), FR: The difference between the maximum and minimum numbers of items processed (distractibility) and PR: TN-E score percentile rank percentage score .

ELIGIBILITY:
Inclusion Criteria:

* Being an emergency department physician (specialist, intern or practitioner)
* Willingness to participate in the study
* Not being pregnant
* Age over 18 and under 60
* Working in the emergency department for at least 1 year

Exclusion Criteria:

* Being left-handed
* Consumption of coffee or alcohol in the previous 24 hours
* Pregnancy
* History of substance misuse or addiction
* Using medication due to psychiatric disease or sleep disorder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-15 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
The change of attention levels | Change from baseline and 15 minutes after exposure
  Determination of the acute effects of electromagnetic waves (EMW) on the attention levels and concentration of emergency physicians after 15-min cell phone use using the d2 test of attention

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Background] Xu F, Bai Q, Zhou K, Ma L, Duan J, Zhuang F, Xie C, Li W, Zou P, Zhu C. Age-dependent acute interference with stem and progenitor cell proliferation in the hippocampus after exposure to 1800 MHz electromagnetic radiation. Electromagn Biol Med. 2017;36(2):158-166. doi: 10.1080/15368378.2016.1233886. Epub 2016 Oct 3. PMID 27696902
- [Background] El-Gohary OA, Said MA. Effect of electromagnetic waves from mobile phone on immune status of male rats: possible protective role of vitamin D. Can J Physiol Pharmacol. 2017 Feb;95(2):151-156. doi: 10.1139/cjpp-2016-0218. Epub 2016 Sep 5. PMID 27901344
- [Background] Al-Serori H, Kundi M, Ferk F, Misik M, Nersesyan A, Murbach M, Lah TT, Knasmuller S. Evaluation of the potential of mobile phone specific electromagnetic fields (UMTS) to produce micronuclei in human glioblastoma cell lines. Toxicol In Vitro. 2017 Apr;40:264-271. doi: 10.1016/j.tiv.2017.01.012. Epub 2017 Jan 24. PMID 28126644
- [Background] Pall ML. Microwave frequency electromagnetic fields (EMFs) produce widespread neuropsychiatric effects including depression. J Chem Neuroanat. 2016 Sep;75(Pt B):43-51. doi: 10.1016/j.jchemneu.2015.08.001. Epub 2015 Aug 21. PMID 26300312
- [Background] Byun YH, Ha M, Kwon HJ, Hong YC, Leem JH, Sakong J, Kim SY, Lee CG, Kang D, Choi HD, Kim N. Mobile phone use, blood lead levels, and attention deficit hyperactivity symptoms in children: a longitudinal study. PLoS One. 2013;8(3):e59742. doi: 10.1371/journal.pone.0059742. Epub 2013 Mar 21. PMID 23555766